CLINICAL TRIAL: NCT06891716
Title: Phase 1 Study to Evaluate [18F]ACI-19626 as a Potential PET Radioligand for Imaging TDP-43 Inclusions in the Brain of Patients With Suspected TDP-43 Proteinopathies Compared With Healthy Controls
Brief Title: [18F]ACI-19626 PET in TDP-43 Proteinopathies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: AC Immune SA (Industry)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACI-19626-FTD-2301; 2024-513097-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Frontotemporal Dementia (FTD); Amyotrophic Lateral Sclerosis (ALS); TDP-43 Proteinopathies; Suspected Limbic Predominant Age-related TDP-43 Encephalopathy (LATE); Alzheimer's Disease (AD)
MeSH Terms: conditions — Frontotemporal Dementia; Amyotrophic Lateral Sclerosis; TDP-43 Proteinopathies; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with suspected TDP-43 proteinopathies (Experimental): The study population will be composed of participants with suspected TDP-43 proteinopathies
  Interventions: Other: [18F]ACI-19626
- Healthy controls (Active Comparator): The study population will be composed of healthy controls.
  Interventions: Other: [18F]ACI-19626

INTERVENTIONS:
Other: [18F]ACI-19626 — [18F]ACI-19626 is an intravenously administered radioactive imaging agent being studied as a potential positron emitting radiopharmaceutical for in vivo imaging of TDP-43 deposits.

SUMMARY:
The goal of this clinical trial is to test whether we can reliably and safely measure the accumulation of pathological protein TDP-43 [involved in rare forms of dementia such as frontotemporal dementia (FTD) and in amyotrophic lateral sclerosis (ALS)] using a new positron emission tomography (PET) tracer called [18F]ACI-19626. Both healthy people and people with (suspected) TDP-43 accumulation will participate to this trial.

The main questions it aims to answer are:

* whether [18F]ACI-19626 is safe and well tolerated when injected into participants
* whether [18F]ACI-19626 reliably detects abnormal TDP-43 in the brain using PET technique.
* whether there are differences in the amount of this protein between people with diseases related to TDP-43 accumulation in the brain and people without these diseases.

Participants will:

* Visit the clinic to consent to their participation and to ensure they are eligible (physical and neurological examinations, questionnaires, blood and urine tests, ECG and MRI in some cases).
* Visit the clinic to receive the tracer [18F]ACI-19626 intravenously and be scanned in a PET scanner, during which blood will be collected.
* Receive a phone call from the clinic 2 to 4 days after the PET scan to report any symptoms and side-effects that they may be having.

Some of the participants may be asked to come again to the clinic for a second PET scan, allowing the researchers to determine if the measurements with the first PET scan are stable and reproducible.

DETAILED DESCRIPTION:
This trial aims to evaluate the effects (i.e. safety and uptake) of a new radiotracer molecule. Study participants will take part in the study by attending two to three study visits over a period of up to 3 months (from the screening visit up to the last study visit).

The study consists of three parts in which a total of up to 45 participants may be included:

Part 1 may include in total up to 15 participants:

* up to 5 healthy controls (HCs)
* up to 5 symptomatic progranulin gene (GRN) and up to 5 symptomatic chromosome 9 open reading frame 72 (C9orf72) mutation carriers with FTD (including prodromal) either with or without motor neuron disease (MND) characteristics.

If the safety and dosimetry are satisfactory in the first subjects and sufficient data are obtained from this part, Part 2 may be initiated.

Part 2 may include in total up to 30 participants including:

* up to 25 patients with TDP-43 proteinopathies: up to 10 additional mutation carriers (including other mutations than GRN and C9orf72, and/or asymptomatic carriers) with FTD (including prodromal) either with or without MND characteristics; up to 10 sporadic or genetic (excluding mutations with known absence of TDP-43 pathology, e.g. Superoxide Dismutase 1 (SOD1) or fused in sarcoma protein gene (FUS)) ALS; up to 10 suspected TDP-43 related sporadic FTD or FTD-MND; up to 5 patients with other neurodegenerative diseases, e.g. AD or suspected Limbic-Predominant Age-related TDP-43 Encephalopathy (LATE) pathology
* up to 5 additional HVs may also be imaged, if necessary, to enable a better distinction of brain binding in this population compared to the population of subjects with TDP-43 proteinopathies

Part 3 aims to assess test-retest reliability. Up to 5 participants from Part 1 and/or Part 2 will have an additional scan within 1 month after their first scan to determine test-retest reliability.

ELIGIBILITY:
Inclusion Criteria for all Participants:

* Subject is able to provide written informed consent (IC), which must be obtained before any assessment is performed.
* Female subjects must not be of childbearing potential, or if they are of childbearing potential to agree to use reliable contraception method(s) and not donate eggs for 30 days after the PET scan. Subjects without documentation of non-childbearing potential will perform serum pregnancy testing at screening and urine pregnancy test before the PET scan. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the PI (e.g., Müllerian agenesis). Women of childbearing potential must commit to remain abstinent (refrain from heterosexual intercourse) or use a reliable form of birth control (e.g. a barrier, hormonal contraception method or intrauterine device), during the study and until 30 days after the last PET scan. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. Women of childbearing potential must commit to not donate ovum during the study and until 30 days after the last PET scan.
* Male subjects with their partners of childbearing potential must commit to the use of a barrier method of contraception during the study and until 90 days after the last PET scan.
* Male subjects must commit to not donate sperm during the study and until 90 days after the last PET scan.
* Willing and able to cooperate with study procedures.
* Ability to tolerate lying in the scanner for up to 90 minutes without excessive movements sufficient to cause significant motion artifact on the PET scans, or if necessary up to 120 minutes with a break.
* For subjects receiving arterial cannulation, adequate circulation to the hand for safe placement of arterial line and coagulation (International Normalized Ratio [INR], Prothrombin Time [PT] and Partial Thromboplastin Time [PTT]).

Additional Inclusion Criteria for Healthy Controls:

* Males and females aged 40-70 years.
* Healthy with no clinically relevant finding on physical and neurological examination at Screening and upon reporting to the clinic for the [18F]ACI-19626 Imaging Visit.
* No family history of TDP-43 proteinopathies, including FTD, ALS, or other early-onset neurological disease associated with dementia and/or movement disorders.
* No personal history of clinically significant neurological and/or psychiatric disorders.
* No evidence of neurodegeneration or other neurological pathology on magnetic resonance imaging (MRI) performed either as part of Screening or on previously acquired MRI scan (within 6 months prior to signing consent).
* Montreal Cognitive Assessment (MoCA) score ≥ 26.
* No cognitive or behavioural impairment as judged by the PI.

Additional Inclusion Criteria for Participants with TDP-43 proteinopathies:

* Males and females aged ≥ 40 years.
* Subjects diagnosed with any of the following: GRN, C9Orf72 or other mutation carriers with the CDR® plus NACC FTLD-GS of ≥ 0.5; sporadic probable behavioral FTD per International consensus criteria or primary progressive aphasia, with or without clinical or electrophysiological indications of MND; ALS meeting the El Escorial criteria of probable or possible ALS; Other neurodegenerative diseases, e.g. AD or suspected LATE pathology
* Confirmed genetic status for the subjects with genetic FTD, FTD-MND or ALS (e.g. GRN, C9orf72 or other mutations)
* For sporadic FTD / FTD-MND subjects: brain MRI consistent with a diagnosis of FTD, with no evidence of focal disease to account for the subject's neurological, cognitive or behavioral symptoms.

Exclusion Criteria for All Participants:

* Current or prior history of any alcohol or drug abuse in the past 2 years.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical condition.
* Known history of hypersensitivity, including hypersensitivity to the active substances used for [18F]ACI-19626 or derivatives, or to any of the associated excipients.
* Prior participation in other research protocols or clinical care during the past year that would result in radiation exposure to an effective radiation dose exceeding the acceptable annual limit (including the procedures in this clinical protocol).
* Pregnant or lactating.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
* Treatment with any antihemostasis medication (e.g., warfarin, heparin, thrombin inhibitors, Factor Xa inhibitors, streptokinase, urokinase, tissue plasminogen activators) within 2 weeks of the planned arterial cannula placement (if performed) of either the baseline or retest imaging.
* Anaemia (for subjects undergoing arterial cannulation) considered clinically significant by the PI
* Coagulopathies
* Loss or donation of blood over 500 mL within four months prior to study visits for subjects undergoing arterial cannulation
* Subject has received an investigational drug within the last 30 days or 5 half-lives prior to the screening assessments, whichever is longer unless there is documented evidence that the subject was treated with placebo only.

Additional Exclusion Criteria for Participants with TDP-43 proteinopathies:

* Prior participation in DMT clinical trials which could interfere with the TDP-43 protein itself or its metabolism, including but not limited to gene therapy, unless there is documented evidence that the subject was treated with placebo only.
* MRI scan showing structural evidence of alternative pathology not consistent with TDP-43 proteinopathies which could cause the subject's symptoms.
* Mutations with known absence of TDP-43 pathology, e.g. SOD1 or FUS.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) assessed by severity (mild, moderate or severe) and causal relationship (unrelated, unlikely, possibly or probably related) | From Informed Consent Signature (screening) to safety phone call after PET scan (i.e. up to 3 months in total)
Number of participants with clinically significant changes in vital signs measurements | During PET scan visit (i.e. at Day 0): before [18F]ACI-19626 injection and after the PET scan is completed
  Vital signs measurements will be performed after the PET scan is completed and will be compared with measurements performed before the injection of [18F]ACI-19626.
Brain uptake of the tracer [18F]ACI-19626 | At the time of the [18F]ACI-19626 PET scan (i.e. at Day 0): 0-90 minutes after injection
  [18F]ACI-19626 brain uptake in relevant regions of interest of the brain will be measured with PET scan and the mean of each group (participants with TDP-proteinopathies and healthy controls) will be calculated.
Assessment of the optimal kinetic model quantification of [18F]ACI-19626 tracer uptake | At the time of the [18F]ACI-19626 PET scan (i.e. at Day 0): 0-90 minutes after injection
  The selection of the optimal kinetic model will be done based on the Akaike's information criterion
Radiation dosimetry after one [18F]ACI-19626 PET scan | At the time of the [18F]ACI-19626 PET scan (i.e. at Day 0): 0-90 minutes after injection
  The radiation dose absorbed by relevant vital organs and the total effective dose will be measured, and the mean of scanned participants will be calculated

SECONDARY OUTCOMES:
Assessment of simplified methods to quantify brain uptake of the tracer [18F]ACI-19626 | At the time of the [18F]ACI-19626 PET scan (i.e. at Day 0): 0-90 minutes after injection
  The validity of simplified reference tissue models will be assessed by determining correlation coefficients with corresponding outcome parameters from the optimal tracer full kinetic model
Variability of the tracer brain uptake between two [18F]ACI-19626 PET scans (test/retest) | At the first [18F]ACI-19626 PET scan and the second [18F]ACI-19626 PET scan (i.e. up to 1 month)
  The repeatability/reliability of the [18F]ACI-19626 brain uptake measures will be assessed by calculating the variability (percentage difference) of the tracer brain uptake between the first and the second [18F]ACI-19626 PET scan for each participant in study Part 3, and the mean will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Elsmarieke van de Giessen, MD, Principal Investigator — Amsterdam UMC; Clinical Lead, Study Director — AC Immune SA
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided